CLINICAL TRIAL: NCT00334477
Title: Efficacy and Safety of Tadalafil 20mg for the Treatment of Erectile Dysfunction in Chronic Renal Patients in Hemodialysis.
Brief Title: Efficacy and Safety of Tadalafil in Hemodialysis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: acbc01
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2006-04

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; chronic renal dysfunction; tadalafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil

SUMMARY:
The purpose of this study is to check the safety and efficacy of a pde5 inhibitor, tadalafil, is a special group of patients: Renal chronic patients in hemodialysis treatment.

DETAILED DESCRIPTION:
In our country, the number of patients in hemodialysis for the treatment of renal chronic dysfunction is very huge. As we know this group has a greater prevalence of sexual dysfunction than the general population, and among these dysfunctions erectile disfunction(ED) occupies maybe the most important position.

With the advent of the increase aging of the nation´s population and the small number of organ donations, the number of men suffering from ED in hemodialysis surely will be very significant causing a very important problem for our health system.

Up to now there´s little indexed publications supporting the use of tadalafil in this special group of men. Another PDE 5 inhibitor, sildenafil, was used in this patients with success and safety but obviously we need other options with the same efficacy.

We intend this study to give us more background to treat ED in this already unfortunate ones.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 70 years old
* Diagnosticated ED for 6 months at least
* Accept the protocol
* Sign the informed consent
* Renal chronic patients in hemodyalisis

Exclusion Criteria:

* History of another PDE5 inhibittor use.
* C.C.I. grade III (NYHA)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
IIEF 5

SECONDARY OUTCOMES:
adverse effects reported

CONTACTS AND LOCATIONS:
Overall Officials: bruno sp carvalho, md, Principal Investigator — University of Pernambuco
Locations (1):
- Hospital de Aeronautica de Recife, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] McMahon C. Efficacy and safety of daily tadalafil in men with erectile dysfunction previously unresponsive to on-demand tadalafil. J Sex Med. 2004 Nov;1(3):292-300. doi: 10.1111/j.1743-6109.04042.x. PMID 16422959
- [Background] McMahon C. Comparison of efficacy, safety, and tolerability of on-demand tadalafil and daily dosed tadalafil for the treatment of erectile dysfunction. J Sex Med. 2005 May;2(3):415-25; discussion 425-7. doi: 10.1111/j.1743-6109.2005.20360.x. PMID 16422874
- [Background] Lewis RW, Sadovsky R, Eardley I, O'Leary M, Seftel A, Wang WC, Shen W, Walker DJ, Wong DG, Ahuja S. The efficacy of tadalafil in clinical populations. J Sex Med. 2005 Jul;2(4):517-31. doi: 10.1111/j.1743-6109.2005.00068.x. PMID 16422847
- [Background] Moore RA, Derry S, McQuay HJ. Indirect comparison of interventions using published randomised trials: systematic review of PDE-5 inhibitors for erectile dysfunction. BMC Urol. 2005 Dec 14;5:18. doi: 10.1186/1471-2490-5-18. PMID 16354303
- [Background] Rosen RC, Shabsigh R, Kuritzky L, Wang WC, Sides GD. The efficacy of tadalafil in improving sexual satisfaction and overall satisfaction in men with mild, moderate, and severe erectile dysfunction: a retrospective pooled analysis of data from randomized, placebo-controlled clinical trials. Curr Med Res Opin. 2005 Nov;21(11):1701-9. doi: 10.1185/030079905X65538. PMID 16307689
- See also: International Society for Sexual Medicine — http://www.issm.info